CLINICAL TRIAL: NCT06309784
Title: Development of a Drill Guidance System to Aid Intra-operative Surgical Drilling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: University of Bath (Other); Great Western Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD 2595; NIHR II-LA-1116-20004 (Other Grant/Funding Number: NIHR)
Record Dates: First submitted 2024-02-09; First posted 2024-03-13 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-02

CONDITIONS: Orthopaedic Surgery
Keywords: orthopaedic; fracture; drill; screw; wire; accuracy
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Participants undergoing orthopaedic Surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drill Guidance System (Experimental): Using a camera based system attached to a standard surgical drill the operating surgeon will use the DGS to drill with the aim of making the drilling more accurate.
  Interventions: Procedure: Drill Guidance System (DGS)

INTERVENTIONS:
Procedure: Drill Guidance System (DGS) — During a standard surgical procedure where a drill/k wire is being inserted the surgeon may choose (in advance) to supplement their drilling with use of the Drill Guidance System. This will be a supplement to normal practice. it is anticipated it will make surgery more accurate, swifter and safer. If however the surgeon is not finding the DGS useful it can be abandoned and standard drilling with X-ray guidance used

SUMMARY:
The Investigators have developed a camera based drill guidance system to improve the accuracy of surgical drilling. The aim of the study is to assess:

Accuracy in vivo Safety Acceptability of use amongst surgeons and theatre staff

DETAILED DESCRIPTION:
This project is a collaboration between the Royal United Hospitals Bath and the Department of Mechanical Engineering at the University of Bath in the development of a drill guidance system to aid intra-operative surgical drilling in Orthopaedic and trauma surgery. The types of operation will include drilling into bones to place screws or wires to develop a track for passage of a screw, suture or other material. The project has been funded by an National Institute for Health Invention for Innovation Grant (NIHR i4i) over 3 years.

The Drill Guide System (DGS) has been developed so it can be attached to a surgical drill with the overall aim of improving the accuracy of surgical drilling of holes in bones. The drilling will be performed as standard, i.e. as required for any specific operation. The drill guide will be an adjunct to visual observation by the surgeon and fluoroscopy (peri-operative radiographs - X-rays). The surgeon can decide to not use the drill guide if it is considered to be hampering the operation. A camera and computer based system attached to a surgical drill will be used to improve drilling accuracy in an operating theatre

The Drill Guidance system has undergone rigorous testing and various laboratory trials with surgeons and operating staff as part of development of the design.

The final prototype will be used as part of a wider clinical trial involving Orthopaedic Surgeons at the Royal United Hospitals Bath and the Great Western Hospital, Swindon (within the NHS) to test the efficacy and value of the system during surgery.

The Investigators intend to recruit up to 30 surgical patients as part of the trial from two sites.

Background: It is recognised clinically and in laboratory studies that "freehand" drilling has appreciable inaccuracies. This risks misplacement of screws potentially compromising surgical outcome and increasing the risk of complications.

Furthermore, inaccurate initial drilling can lead to inaccurate subsequent drilling and so suboptimal positioning of the screw/wire with potential adverse outcomes and increased costs. The screw may be placed and then have to be changed. A new different length screw may be required with the first screw discarded with further costs.

ELIGIBILITY:
Inclusion Criteria:

* adults, i.e. 18 years or over;
* awaiting orthopaedic or trauma surgery;
* have capacity to consent to participate in the study
* the proposed operation is deemed to be appropriate by the treating Orthopaedic surgeon for use of the DGS

Exclusion Criteria:

* children, i.e. < 18 years of age
* the patient is unable to give informed consent;
* the surgeon does not feel able to use the DGS
* the surgeon does not feel use of the DGS is appropriate for the type of surgery required

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of placement of a screw or K wire in scaphoid bones | 3 months
  1.Scaphoid fractures: "best practice" is screw placement in the central third of the scaphoid. This has been defined using CT scans in the Scaphoid Waist Internal Fixation for Fractures (SWIFFT) trial. When fixing a scaphoid fracture the surgeon will aim to place the screw in the central third of the scaphoid (standard) unless otherwise recorded. The screw position will be measured as central or off-centre (as in SWIFFT trial). The data from the SWIFFT trial will be used as a benchmark
  Measurements will be made with the computer measuring system on the Patient Archiving Communication System
Accuracy of placement of a screw or K wire in other bones | 3 months
  Other fractures: at the point the surgeon plans to drill for the material screw/wire they will declare the planned exit point of the screw/wire using x and y co-ordinates in mm relative to a defined bony landmark prior to the use of the Drill Guide System. The screw/wire position on post-operative CT scans will be defined by the position of the tip of the screw/wire (or its projection to the outer cortex of the bone if it does not reach). This will be compared to the planned exit point to give distance and vector measurements
  Measurements will be made with the computer measuring system on the Patient Archiving Communication System

SECONDARY OUTCOMES:
Length of material part of the procedure | Duration of the operation
  The length of time performing the part of the surgical procedure when the DGS is used. There are no baseline data against which to compare. This should give an indicator of speed/ease of use.
Number of fluoroscopy (perioperative X-ray) images performed | Duration of the operation
  The number of fluoroscopy images performed peri-operatively whilst using DGS; for scaphoid fractures data will be compared with data from > 200 equivalent operations in the Scaphoid Waist internal fixation for fractures (SWIFFT) trial. For other operations the number of images taken when using the DGS will be recorded. There are no baseline data but the data can be used as an estimate of ease of use
Number of patients with treatment related adverse events as assessed by CTCAE v4.0 | WIthin 3 months of surgery (the planned follow-up period)
  The key adverse events we will review:
  Screw misplacement (prime complication).
  * scaphoid fractures: when the screw is not in the central third of the scaphoid
  * other operations: when the screw/wire tip (or its projection to the outer cortex of the bone) is outside the chosen limits - 2mm in either plane at a distance of 30mm.
  Bone: Fracture mal-alignment post-operatively as shown on the initial post-operative radiographs and any subsequent radiographs/scans.
  Soft tissue: Possible soft tissue complications e.g. infection, and nerve and tendon injury, will be sought and recorded in the clinical notes at each standard clinical appointment
Immediate acceptability to surgeons and theatre staff | 3 months, i.e. duration of the study
  Following consent the surgeons and theatre staff will be asked to complete a short questionnaire after each operation.
Initial acceptability to surgeons and theatre staff | 3 months, i.e. duration of the study
  After the first 5 operations there will also be a debrief in person to get immediate feedback
Overall acceptability to surgeons and theatre staff | 3 months
  Qualitative data will be collected via two focus groups held either face to face at each site or via Teams to include surgeons and theatre staff. These will collect user views on ease of use, problems encountered and areas for improvement. The focus groups will be recorded to allow for transcription and analysis of themes after all participants have completed their initial operation. Attendance at these focus groups will be optional for theatre staff and consent will be sought

CONTACTS AND LOCATIONS:
Overall Officials: Adam Smith, FRCS (T and O), Principal Investigator — Great Western Hospitals NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Royal United hospitals NHS Foundation Trust, Bath
  - Great Western Hospital MHS foundation Trust, Swindon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langeveld ARJ, Rustenburg CME, Hoozemans MJM, Burger BJ, Meuffels DE. To Improve Your Surgical Drilling Skills, Make Use of Your Index Fingers. Clin Orthop Relat Res. 2019 Jan;477(1):232-239. doi: 10.1097/CORR.0000000000000557. PMID 30394951
- [Background] Brioschi V, Cook J, Arthurs GI. Can a surgeon drill accurately at a specified angle? Vet Rec Open. 2016 Jul 14;3(1):e000172. doi: 10.1136/vetreco-2016-000172. eCollection 2016. PMID 27547423
- [Result] Dias JJ, Brealey SD, Fairhurst C, Amirfeyz R, Bhowal B, Blewitt N, Brewster M, Brown D, Choudhary S, Coapes C, Cook L, Costa M, Davis T, Di Mascio L, Giddins G, Hedley H, Hewitt C, Hinde S, Hobby J, Hodgson S, Jefferson L, Jeyapalan K, Johnston P, Jones J, Keding A, Leighton P, Logan A, Mason W, McAndrew A, McNab I, Muir L, Nicholl J, Northgraves M, Palmer J, Poulter R, Rahimtoola Z, Rangan A, Richards S, Richardson G, Stuart P, Taub N, Tavakkolizadeh A, Tew G, Thompson J, Torgerson D, Warwick D. Surgery versus cast immobilisation for adults with a bicortical fracture of the scaphoid waist (SWIFFT): a pragmatic, multicentre, open-label, randomised superiority trial. Lancet. 2020 Aug 8;396(10248):390-401. doi: 10.1016/S0140-6736(20)30931-4. PMID 32771106